CLINICAL TRIAL: NCT02562963
Title: Phase 1/2 Study of Natural Killer T Cell Infusion in Patients With Advanced Solid Tumor
Brief Title: Clinical Efficacy and Safety of NKT Cell Infusion in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minghui Zhang (Other)
Collaborators: Shanghai Public Health Clinical Center (Other Government); First Hospital of Tsinghua University (Other)
Responsible Party: Sponsor-Investigator, Minghui Zhang, Associate Professor, Tsinghua University
Organization: Tsinghua University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKT-THU2015; SHAPHC-CA-150209 (Other: Shanghai Public Health Clinical Center); BHXH-CA-150413 (Other: Hua Xin Hosptial First Hosptial of Tsinghua University)
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer; Gastric Cancer; Hepatocellular Carcinoma; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Carcinoma, Hepatocellular; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- natural killer T cell (Experimental): The eligible patients are infused with two doses of (4±0.5)x10^9 NKT cells in one course of treatment. Intervention: Biological: NKT cell
  Interventions: Biological: natural killer T cell

INTERVENTIONS:
Biological: natural killer T cell — The eligible patients are infused with two doses of (4±0.5)x10^9 NKT cells in one course of treatment.

SUMMARY:
Natural killer T (NKT) cells are a unique subset of lymphocytes that present a mixed T-NK phenotype. Our hypothesis is that Natural killer T cells may decrease the tumor burden and improve overall survival. The purpose of this study is to determine whether Natural killer T (NKT) cells are effective and safe in the treatment of patients with unresectable advanced solid tumor.

DETAILED DESCRIPTION:
According to the Annual Report of Cancer Registration in China 2014, lung cancer, gastric cancer, liver cancer and colorectal cancer have become the top 4 solid tumors with the highest morbidity and mortality rates. So far, the main treatment modalities for these tumors have been surgery, radiotherapy and chemotherapy. However, the effect of conventional therapy on advanced cancer is limited, tumor metastasis is the major cause of death in patients with advanced cancer. With the development of oncology and immunology in recent years, immunotherapy represents a novel path to obtain a durable and long-lasting response in cancer patients.

Natural killer T (NKT) cells are a unique subset of lymphocytes that present a mixed T-NK phenotype. NKT cells are expanded conventionally from peripheral blood mononuclear cells by addition of a variety of cytokines in vitro culture. Our previous studies demonstrated that the expansion of NKT cells in a clinical usage scale from peripheral blood mononuclear cells is feasible. Those expanded NKT cells exhibit antitumor effect in vitro and in vivo (tumor -bearing nude mice) against a variety of tumor cells. Furthermore, intravenous infusion of a single dose of 4X10^9 NKT cells in mice has been proved safe.

The purpose of this study is to evaluate the efficacy and safety of NKT cells in patients with unresectable advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years, Male or Female
* Histological or cytologically diagnosis of advanced non-small cell lung cancer, or advanced gastric cancer, or advanced hepatocellular carcinoma, or advanced colorectal cancer
* Patients' tumor tissue (formalin-fixed, paraffin-embedded) must be sufficient for diagnosis of cancer by a certified Laboratory of Pathology
* Laboratory values within the following ranges prior to receiving treatment of study agent: Hemoglobin≧11.0 g/dL, Neutrophils count≧1.5×l09/L, Lymphocytes count≧lower limit of institutional normal, Platelet count≧80×l09/L, Serum creatinine≦2.0 mg/dL, Serum bilirubin≦2 x upper limit of institutional normal, AST/ALT≦2 x upper limit of institutional normal
* No dyspnea at rest. Oxygen saturation ≥90% on room air
* Able to tolerate apheresis procedure including placement of temporary apheresis catheter
* No genetic disease
* No chemotherapy and radiation therapy to be planned recently
* Fertile females/males must consent to use contraceptives during participation of the trial. Women of child bearing potential must have a negative pregnancy test prior to receiving treatment of study agent within 7 days
* Patients must have a Karnofsky performance status greater than or equal to 80%
* Life expectancy greater than twelve months
* Able and willing to give witnessed, written informed consent form prior to receiving any study related procedure
* Agree that progress of the disease must be radiographically measurable by computerized tomography (CT) scanning technique or magnetic resonance imaging (MRI) (per RECIST1.1 criteria)
* Agrees to participate in long-term follow-up for up to 3 years, if received NKT infusion

Exclusion Criteria:

* Organ dysfunction defined as follows: Significant cardiovascular disease (i.e. New York Heart Association [NYHA] class 3 congestive heart failure, myocardial infarction within the past six months, unstable angina, coronary angioplasty within the past six months, uncontrolled atrial or ventricular cardiac arrhythmias; Child-Pugh C; Renal function failure or uremia; Respiratory failure; Disturbance of consciousness
* Suffering from lymphoma or leukemia
* Serious infections requiring antibiotics, bleeding disorders
* Patients with myelodysplastic syndrome (MDS)
* History of immunodeficiency disease or autoimmune disease
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Known central nervous system tumors including metastatic brain disease, unless treated and stable
* Other malignancy within 3 years prior to entry into the study
* Negative HIV antigen and antibody, Hepatitis B surface antigen and Hepatitis C PCR within 21 days prior to enrollment
* Patients with chronic disease which is undergoing immune reagents or hormone therapy
* Previous bone marrow or stem cell transplant, or organ allograft
* Within concurrent chemotherapy
* Concomitant treatment with corticosteroids (Topical or inhalational corticosteroids are permitted)
* Concurrent other medical condition that would prevent the patient from undergoing protocol-based therapy
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dose of study agent
* Pregnant or breast-feeding patients
* Mental impairment or addictive disorders that may compromise the ability to give informed consent
* Lack of availability of a patient for immunological and clinical follow-up assessment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events following infusion of NKT cells | 30 days post-infusion
  liver dysfunction, kidney dysfunciton, shivering, diarrhea, fever and more
Objective Response Rate (ORR), confirmed by CT or MRI, or confirmed by biopsy | up to 24 weeks
  The proportion of participants with complete remission and partial remission which judged by RECIST v1.1

SECONDARY OUTCOMES:
Hematology | Baseline, 1 day, 7 days, 14 days and 28 days after cell infusion
  Hematology, include erythrocytes, leukocytes, platelets, T lymphocytes, B lymphocytes, Natural killer cell, NKT, CD4/CD8, Th1/Th2, Th17 cell and Treg lymphocytes
Serological analysis | Baseline, 1day, 7 days, 14 days and 28 days after cell infusion
  Serological analysis, include immunoglobulin G, immunoglobulin A, immunoglobulin D, immunoglobulin E and immunoglobulin M. Albumin (ALB), Alanine aminotransferase (ALT), Aspartate Aminotransferase (AST), Prealbumin (PA), total bilirubin (TB), and direct bilirubin (DB); Blood urea nitrogen (BUN), Urea (UA), and Crea (Cr); Total cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), triglycerides (TG), very low density lipoprotein cholesterol (VLDL-C), and Non-HDL-C; blood sugar
Overall Survival (OS) | Approximately 3 years
  The time from the beginning of ransomization to death from any cause
Progression-Free Survival (PFS) | Approximately 1 years
  The time from randomization to the first recording of disease progression (RECIST v1.1)
Tumor Marker | up to 24 weeks
  CEA, AFP and more

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Zhang, PhD, Study Chair — Tsinghua University
Locations (2):
- China (2):
  - Hua Xin Hosptial First Hosptial of Tsinghua University, Beijing
  - Shanghai Public Health Clinical Center, Shanghai

IPD SHARING:
Plan to Share IPD: No